CLINICAL TRIAL: NCT00314483
Title: Evaluation of Potential Mesenchymal Stem Cells for the Treatment of Graft Versus Host Disease Following an Allogeneic Stem Cell Transplant
Brief Title: Evaluation of the Role of Mesenchymal Stem Cells in the Treatment of Graft Versus Host Disease
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Christian Medical College, Vellore, India (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMCMSC_GVHD012006
Record Dates: First submitted 2006-04-12; First posted 2006-04-14 (Estimated); Last update posted 2007-07-06 (Estimated); Status verified 2007-07

CONDITIONS: Graft vs Host Disease
Keywords: Mesenchymal stem cells; GVHD; Treatment; Steroid refractory GVHD
MeSH Terms: conditions — Graft vs Host Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: Mesenchymal Stem Cell Infusion

SUMMARY:
Mesenchymal stem cells (MSC) have been shown to have immunosuppressive properties. Following a bone marrow/peripheral blood stem cell transplant, a proportion of patients develop a condition called 'graft versus host disease' (GVHD). In this condition the transplanted cells recognize the recipient as foreign and bring about an immune-mediated destruction of tissues. The treatment for this condition is to use drugs that will cause immunosuppression. A small subset of these patients develop a severe form of GVHD (Grade III or IV) which, in spite of the best currently available treatment, is associated with eventual death in more than 90% of cases. The investigators propose to use infusions of expanded MSC from the donor to treat this condition. A few reports on this approach have already been published in peer reviewed journals and preliminary results appear to be promising. The investigators are also aware that larger trials have been initiated to study this. After getting written informed consent, the investigators will infuse expanded MSC into patients who develop steroid-resistant GVHD.

DETAILED DESCRIPTION:
A single center non randomized, non blinded Phase I/II clinical trial is proposed to study the role of mesenchymal stem cells (MSC) in the management of steroid refractory graft versus host disease (GVHD) following an allogeneic stem cell transplant.

Patients who develop grade II to IV GVHD following an allogeneic stem cell transplant will be enrolled. MSC will be expanded from the donors of all patients who develop GVHD. Expanded MSC will be infused at a dose of 1-2 million cells/kg in patients who have steroid refractory GVHD.

Response to therapy will be studied using established criteria for grading GVHD.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained from patient and donor
* Any patient who has undergone HLA-matched related allogeneic stem cell transplantation with steroid refractory Grades II-IV acute GVHD
* Prednisolone 2 mg/kg/day (or equivalent doses of methylprednisolone, etc.) for at least one week

Exclusion Criteria:

* Invasive fungal disease
* Active cytomegalovirus (CMV)/Epstein-Barr virus (EBV)/varicella disease
* Relapsed malignancy

Ages: 2 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 25 (Estimated)
Dates: Start 2007-06; Study Completion 2008-06 (Estimated)

PRIMARY OUTCOMES:
Control of GVHD | 8 weeks

SECONDARY OUTCOMES:
Infusional toxicity | 48 hours
Risk of relapse | One year

CONTACTS AND LOCATIONS:
Overall Officials: Vikram Mathews, MD, Principal Investigator — Christian Medical College, Vellore, India
Locations (1):
- Department of Haematology, Christian Medical College, Vellore, Tamil Nadu, India